CLINICAL TRIAL: NCT01148693
Title: Comparing Addition of Gentamicin vs. Placebo in Preventing Post ERCP Cholangitis in Non-calculus Stenting
Brief Title: Gentamicin in Preventing Post Endoscopic Retrograde Cholangiopancreatography (ERCP) Cholangitis in Non-calculus Stenting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Norouzi, gastroenterology fellow in DDRC, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DDRC-88/19
Record Dates: First submitted 2010-06-19; First posted 2010-06-22 (Estimated); Results first posted 2011-08-22 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-07

CONDITIONS: Cholangitis
Keywords: Cholangitis; Cholangiopancreatography, Endoscopic Retrograde; stents; cholestasis
MeSH Terms: conditions — Cholangitis; Cholestasis | interventions — Gentamicins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gentamicin (Active Comparator): adding 10mg gentamicin to every 10 ml of contrast media
  Interventions: Drug: gentamicin
- Placebo (Placebo Comparator): Identical placebo
  Interventions: Drug: gentamicin; Drug: Placebo

INTERVENTIONS:
Drug: gentamicin — 10mg per 10ml of contrast media
  Other Names: Brand name: Gentamicin
Drug: Placebo — Distilled water
  Arms: Placebo

SUMMARY:
Cholangitis is the most prevalent infectious complication of ERCP. Stenting of biliary strictures and stenosis is one of important risk factors for post-ERCP cholangitis. Adding antibiotics to contrast media has proposed in some studies for prevention of cholangitis but remains controversial. In this study we compare effect of adding gentamicin versus placebo in preventing cholangitis in patients who undergone endoscopic stenting for non-calculus strictures and stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-calculus biliary obstruction who need palliative treatment

Exclusion Criteria:

* Fever (> 37.8 Celsius)
* Leukocytosis (WBC > 10,000 /mm3)
* Not candidate for surgical cure of obstruction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rasoul Sotudemanesh, MD, Study Chair — Tehran Medical University of Medical Science associate professor
Locations (1):
- TUMS Digestive Disease Research Center, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Norouzi A, Khatibian M, Afroogh R, Chaharmahali M, Sotoudehmanesh R. The effect of adding gentamicin to contrast media for prevention of cholangitis after biliary stenting for non-calculous biliary obstruction, a randomized controlled trial. Indian J Gastroenterol. 2013 Jan;32(1):18-21. doi: 10.1007/s12664-012-0208-y. Epub 2012 Oct 19. PMID 23081843

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2009 and October 2010 all patients with non-calculus biliary obstructions including cholangiocarcinoma, pancreatic cancer, sclerosing cholangitis, postsurgical benign biliary strictures and biliary stenosis due to metastatic cancers to biliary tree who were candidate for palliative stenting, were included in this study.
Pre-assignment Details: Exclusion criteria were patients with biliary stones, patients who were candidate for surgical cure, and patients who were already febrile.
Groups:
- Gentamicin: participitants for whom gentamicin with a dose of 10mg/10ml was added to contrast media during endoscopic cholangiopancreatography
- Placebo: participitants for whom identical placebo with a dose of 10mg/10ml was added to contrast media during endoscopic cholangiopancreatography
Period: Overall Study
Arm/Group | Gentamicin | Placebo
Started | 70 | 67
Completed | 57 | 57
Not Completed | 13 | 10
Not completed — Attempts for cannulation were failed | 13 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gentamicin | Placebo | Total
Number analyzed (Participants) | 70 | 67 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 39 | 79
  >=65 years | 30 | 28 | 58
Age Continuous [Mean (Standard Deviation); unit: years] | 62.59 (15.082) | 66.74 (14.145) | 64.62 (14.533)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 20 | 48
  Male | 42 | 47 | 89
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 70 | 67 | 137

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cholangitis
Description: After Endoscopic Retrograde CholangioPancreatography (ERCP) in 3 following days we check all participants for syptoms of cholangitis (fever, chills, right upper qudrant (RUQ) pain, leukocytosis) and ruling out other diagnoses than cholangitis
Time Frame: 72 hours
Measure: Number; unit: participants
Groups:
- Gentamicin: patients for whom 10m/10cc of gentamicin is added to contrast during ERCP
- Placebo: patients for whom distilled water is added to contrast during ERCP
Arm/Group | Gentamicin | Placebo
Number analyzed (Participants) | 57 | 57
participants | 5 | 5
Statistical Analysis 1: Comparison: Gentamicin vs Placebo; Null hypothesis: Adding gentamicin to contrast medium during ERCP has no relation with postERCP cholangitis Power calculation: 80%; Test type: Superiority or Other; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Gentamicin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 0/57 | 0/57

LIMITATIONS AND CAVEATS:
No limitation other than small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No